CLINICAL TRIAL: NCT02234401
Title: A Mixed Methods Study Comparing the Clinical Efficacy With the Patient Experience of Non-invasive Ventilation During an Acute Exacerbation Complicated by Respiratory Failure in Adult Cystic Fibrosis
Brief Title: Non Invasive Ventilation for Acute Exacerbations in Adult CF
Acronym: NIVinCF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manchester Metropolitan University (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Susan C Johnson, Consultant Physiotherapist, Manchester Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1199
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Cystic Fibrosis; Respiratory Failure
Keywords: Cystic Fibrosis; Noninvasive ventilation; Non invasive ventilation; Acute respiratory exacerbation; Bi level pressure support
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Insufficiency | interventions — Noninvasive Ventilation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non invasive ventilation (NIV) (Experimental): Non invasive ventilation used for the first 7 days of study
  Interventions: Device: Bi level pressure support
- Standard Care (Active Comparator): High Flow Controlled Oxygen Therapy
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: Bi level pressure support
  Other Names: Noninvasive ventilation; NIV
  Arms: Non invasive ventilation (NIV)
Other: Standard Care
  Arms: Standard Care

SUMMARY:
Cystic Fibrosis (CF) is a life limiting illness. Median predicted UK survival is 41.4 years (UK CF Registry 2011). The commonest cause of death is respiratory failure.

Non invasive ventilation (NIV) is a system which delivers a preset pressure to supplement the size and depth of each breath. It is introduced in CF to manage established respiratory failure. A nose or a mask which covers both the nose and mouth allows flexible ventilation, is used just at night, or for part of the day in addition or for 24 hours as clinical status indicates. It is introduced within a normal ward environment and then continued longterm at home.Once respiratory failure is established longterm noninvasive ventilation is introduced throughout 24 hours and multidisciplinary assessment concludes that the timing is appropriate for the individual.

This study aims to evaluate a potential development of current practice: the use of non invasive ventilation during hospital admission only to enhance recovery from an acute exacerbation which has caused respiratory failure in those individuals where long term non invasive ventilation is not yet indicated. A mixed methods design will allow description of the experience of noninvasive ventilation during a semistructured interview to add to understanding of the results from an experiment designed to measure the differences between noninvasive ventilation and standard care.

Aim: To compare the clinical efficacy with the patient experience of NIV on recovery from an acute respiratory exacerbation complicated by respiratory failure in adult Cystic Fibrosis.

DETAILED DESCRIPTION:
Design: The study will use a mixed methodology and it will be in 2 phases. Phase I A group randomised controlled trial

The following measurements will be performed on days 1, 3, 7, 10, 14 and twice weekly until discharge:

The exact timing of measurements will be planned by the participant and the researcher.

All of the outcome measures form part of routine clinical practice except the symptom score; the Cystic Fibrosis Respiratory Symptoms Diary (CFRSD V2.0) (Goss et al., 2009)

1. Early morning and day time carbon dioxide (CO2) level.
2. Day time oxygen levels
3. Lung function Forced Expiratory Volume in 1 second (FEV1) and Forced Vital Capacity (FVC)
4. Day time resting Respiratory Rate (RR), Heart Rate (HR)
5. Symptom score CFRSD

Phase II A qualitative exploration of the experience of using NIV for adults with Cystic Fibrosis during an acute exacerbation

Methods: Prior to discharge a semistructured interview designed to explore the experience of using noninvasive ventilation will be undertaken by a clinical psychologist from the Cystic Fibrosis multidisciplinary team. The interviews will be undertaken purely for the research project, recorded and transcribed verbatim by the lead investigator. Thematic analysis will be undertaken to interpret and explore the individual's experience. Credibility checking of interpretation will be undertaken by the clinical psychologists and within academic supervision sessions.

ELIGIBILITY:
Inclusion Criteria:

* Adult Cystic Fibrosis
* Hospital admission to Pearce Ward Manchester Adult Cystic Fibrosis Centre
* Acute respiratory exacerbation conforming with a standard definition of pulmonary exacerbation (Fuchs et al 1994).
* An admission day time CO2 > 6 kilopascal (kPa) on standard therapy
* Freely given informed consent.-
* 24.3.15 substantial amendment approval for an admission early morning CO2 > 6 kPa

Exclusion Criteria:

* A day time CO2 >8.0 kPa
* respiratory acidosis
* clinical exclusion by CF consultant physician or clinical psychologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change in day time carbon dioxide (CO2) | Day 7

SECONDARY OUTCOMES:
Early morning oxygen (O2) and CO2 levels | days 1,3,5,7,10 and 14
Lung function (FEV1 and FVC) | Day 7, 14
Respiratory Rate | days 1,3,5,7,10 and 14
Heart Rate | Days 1,3,5,7,10 and 14
Symptom score (CFRSD) | days 1,3,5,7,10 and 14
  Cystic Fibrosis Respiratory Symptom Diary (Daily Recall)

OTHER OUTCOMES:
Semi structured interview | Day 14
  Psychologist delivered semi structured interview discussing participant experience of non invasive ventilation (NIV)

CONTACTS AND LOCATIONS:
Overall Officials: Susan C Johnson, MSC MCSP, Principal Investigator — Manchester Adult Cystic Fibrosis Centre, University Hospitals South Manchester
Locations (1):
- Manchester Adult Cystic Fibrosis Centre, University Hospitals South Manchester, Wythenshawe, Manchester, United Kingdom